CLINICAL TRIAL: NCT04614961
Title: Database Concerning Patients Consulting the Obesity Clinic of University Hospitals Leuven
Brief Title: Database Concerning Patients Consulting the Obesity Clinic
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62590
Record Dates: First submitted 2020-10-05; First posted 2020-11-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity; Bariatric Surgery
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutrition Therapy; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with overweight, obesity or after bariatric surgery: Patients with overweight, obesity or after bariatric surgery
  Interventions: Other: Lifestyle therapy - individual; Other: Lifestyle therapy - group; Other: Medical therapy; Procedure: Bariatric surgery

INTERVENTIONS:
Other: Lifestyle therapy - individual — Individual therapy
Other: Lifestyle therapy - group — Group therapy
Other: Medical therapy — Medical therapy
Procedure: Bariatric surgery — Surgical and endoscopic therapy

SUMMARY:
A registry of individuals that visit the Obesity Clinic of the University Hospitals of Leuven will be established. The objective of this registry is to improve the knowledge about obesity, the treatment of obesity and its outcomes.

DETAILED DESCRIPTION:
A registry/database is constructed with data of the individuals that visit the Obesity Clinic of the University Hospitals of Leuven. Data will be obtained from the screening visits and all follow-up visits in terms of sociodemographics, treatment and treatment outcomes, disease impact, biochemistry, questionnaires, QoL, …

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 years or older
* Subjects with overweight, obesity or after bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with overweight, obesity or after bariatric surgery
Sampling Method: Probability Sample
Enrollment: 999999 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Routine treatment data (sociodemographics, treatment and treatment outcome, disease impact, biochemistry, questionnaires, ...) | up to 100 years
  The objective is to develop an Obesity Clinic registry to collect routine treatment data (sociodemographics, treatment and treatment outcome, disease impact, biochemistry, questionnaires, ...) using the electronic medical record to improve the knowledge on obesity, the treatment of obesity and its outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Obesity Clinic University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided